CLINICAL TRIAL: NCT04897022
Title: Phase I Dose Escalation and Local Control Study of Pembrolizumab + Intensity-Modulated Pleural Radiation Therapy (IMPRINT) for Malignant Pleural Mesothelioma
Brief Title: A Study of Pembrolizumab and Radiation Therapy in People With Mesothelioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-197
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: malignant pleural mesothelioma; MPM; intensity-modulated pleural radiation therapy; IMPRINT; Pembrolizumab; 21-197; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — pembrolizumab; Imprint II

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with malignant pleural mesothelioma (MPM) (Experimental): Participants will be diagnosed with malignant pleural mesothelioma and be deemed unresectable per thoracic surgeon assessment
  Interventions: Drug: Pembrolizumab; Radiation: IMPRINT

INTERVENTIONS:
Drug: Pembrolizumab — Fixed dose of pembrolizumab 200mg IV q3 weeks
Radiation: IMPRINT — The starting radiation dose will consist of 400cGy x5 fractions. Doses will be escalated by 100cGy per fraction (i.e. 400cGy, 500cGy, 600cGy) for a total of 3 dose levels. The MTD will be evaluated using a modified Continuous Reassessment Method. Dose limiting toxicities (DLTs) are defined as any treatment-related non-hematologic toxicity with a CTCAE v5 Grade ≥3 or grade ≥2 pneumonitis that requires use of steroids occurring after the start of IMPRINT through the first 3 months after the last fraction.
  Other Names: intensity-modulated pleural radiation therapy

SUMMARY:
The purpose of this study is to find out whether IMPRINT in combination with pembrolizumab is a safe treatment for people with malignant pleural mesothelioma (MPM).The highest dose of IMPRINT that causes few or mild side effects when given in combination with pembrolizumab will be found. Once the highest safe dose of IMPRINT is found, it will be tested in combination with pembrolizumab in future participants to see whether the combination may be an effective treatment for MPM.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of malignant pleural mesothelioma
* Unresectable per thoracic surgeon assessment
* At least one prior line of systemic therapy. Note: Patients who were on prior immunotherapy are eligible.
* ECOG 0-1
* PFTs: DLCO >40% predicted, FEV1 >50% predicted
* Male/female participants who are at least 18 years of age on the day of signing informed consent
* Disease outside the ipsilateral thorax allowed as long as it has either been treated definitively and been stable for 6 months

Male participants:

* A male participant must agree to use a contraception as detailed in Appendix 1 of this protocol during the treatment period and for at least 30 days, corresponding to time needed to eliminate any study treatment(s) (pembrolizumab and or any active comparator/combination) plus an additional 120 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose after the last dose of study treatment and refrain from donating sperm during this period.

Female participants:

* A female participant is eligible to participate if she is not pregnant (see Appendix 1), not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 1 OR
  2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 1 during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatment(s) (pembrolizumab and or any active comparator/combination) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment.
* The participant (or legally authorized representative if applicable) provides written informed consent for the trial.
* Have a ECOG performance status of 0 to 1. Evaluation of ECOG is to be performed within 30 days prior to the date of allocation.
* Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 45 days prior to the start of study treatment.

Table 1: Adequate Organ Function Laboratory Values

System: Hematological Absolute neutrophil count (ANC) ≥ 1.5 K/mcL Platelets ≥ 100 K/mcL Hemoglobin ≥ 9.0 g/dL

System: Renal Creatinine OR Measured or calculated^b creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤ 1.5 x ULN OR ≥ 30 mL/min for participant with creatinine levels >1.5 x institutional ULN

System: Hepatic Total bilirubin: ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5 x ULN AST (SGOT) and ALT (SGPT): ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastases)

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

^b: Creatinine clearance (CrCl) should be calculated per institutional standard.

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

* Newly diagnosed MPM
* Prior thoracic radiation therapy or intrapleural therapy
* Bulky disease in the fissure preventing IMPRINT
* Serious infection, concurrent active malignancies, or other serious medical illness
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137) within 4 weeks prior to study Day 1 or has not recovered (i.e., ≥ Grade 1 at baseline) from adverse events due to a previously administered agent
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Low grade malignancies not requiring active treatment are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression, clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has undergone major surgery <4 weeks from starting pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of IMPRINT | 6 months
  The first primary objective of this study is to determine the MTD of IMPRINT among the three candidate doses: 400cGy x5 fractions, 500cGy x5 fractions and 600cGy x5 fractions. These dose levels will be evaluated using a modified Continuous Reassessment Method (CRM) starting with the lowest dose level 400cGy x5 fractions. Determined by the first 12 participants enrolled to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Simone, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org